CLINICAL TRIAL: NCT02617524
Title: A Prospective, Open-label Study to Evaluate the Feasibility and Safety of the Valve Medical Dedicated Sheath During Balloon Aortic Valvuloplasty
Brief Title: Dedicated Sheath Feasibility Study
Acronym: BAV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valve Medical (Industry)
Collaborators: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLICL 01446
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Aortic Stenosis
Keywords: dedicated sheath
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valve Medical Dedicated Sheath (Experimental): Valve Medical Dedicated Sheath version 00
  Interventions: Device: Valve Medical Dedicated Sheath version 00

INTERVENTIONS:
Device: Valve Medical Dedicated Sheath version 00 — The Valve Medical Dedicated Sheath is intended to be used as an introducer sheath during BAV procedures

SUMMARY:
Dedicated Sheath feasibility study: A prospective, open-label study to evaluate the feasibility and safety of the Valve Medical Dedicated Sheath during Balloon Aortic Valvuloplasty (BAV).

DETAILED DESCRIPTION:
This is an open-label, prospective, single arm clinical study. Up to 15 patients undergoing valvular intervention will be enrolled. Follow up will take place at 1, 6 and 24 hours post procedure. No follow up visits are required.

During the study, the patient will undergo the following tests:

* Physical examination (includes blood pressure, age, height, weight).
* Echo assessments prior to procedure.
* Hemodynamic study prior and post BAV.
* Full blood count
* Angiography

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient understands the implications of participating in the study and provides written informed consent.
* The patient has an indication for balloon aortic valvuloplasty (BAV).

Exclusion Criteria:

* Peripheral vessel anatomy or peripheral vascular disease that would preclude the insertion of the 12 Fr. sheath.
* Any illness or condition which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Device success | Outcome measures will be assessed at 1, 6 and 24 hours post procedure.
Procedure Safety: Adverse Event Assessment for device related and unrelated events | Outcome measures will be assessed at enrollment, throughout the procedure and 1, 6 and 24 hours post procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel